CLINICAL TRIAL: NCT04273386
Title: Mouth Handicap in Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tugba Civi Karaaslan, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ISTANBULC1
Record Dates: First submitted 2019-11-26; First posted 2020-02-18 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Scleroderma; Systemic Sclerosis; Mouth Diseases
Keywords: Scleroderma; Systemic sclerosis; Mouth
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic; Mouth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation (Experimental): Cases will be evaluated for oral health and data will be recorded.
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — The study will be carried out with the method of filling the evaluation form which is printed on paper with ballpoint pen.

SUMMARY:
In this study, it is aimed to investigate the mouth handicap in Systemic Sclerosis.

DETAILED DESCRIPTION:
Systemic Sclerosis is an autoimmune connective tissue disease with fibrosis. Although its etiology and pathogenesis have not been clearly defined, it has a chronic course. Systemic sclerosis is estimated to affect approximately 300,000 people in the United States. Most commonly, it affects adults and women.

Narrowing of the mouth opening and mouth pain are the two most important causes reported by adults with systemic sclerosis. In patients with systemic sclerosis, orofacial findings such as microstomy or reduced mouth opening are frequently seen. Microstomy is defined as the distance between the incisors is less than 40 millimeters. In severe microstomy, this distance is less than 30 millimeters. It is approximately 33 millimeters in adults with systemic sclerosis. Microstomy in systemic sclerosis mainly results from submucosal collagen deposits that contribute to fibrosis in the perioral tissue. Microstomy is seen in 43% to 80% of adults with systemic sclerosis.

When the current literature is examined, Bongi et al. evaluated the effectiveness of face-specific programs, which are applied together with general rehabilitation programs in patients with systemic sclerosis; they demonstrated that these techniques improve disability, health-related quality of life (HRQoL), and facial functionality.

In this study, it is aimed to investigate the mouth handicap in Systemic Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with systemic sclerosis
* Stability of medical treatments
* Turkish literacy

Exclusion Criteria:

* The patient has a history of neurological disease or trauma that may affect his symptoms
* Oral treatment for the last 6 months
* Being in active phase of the disease
* Skin infection and presence of open wound
* Having used dental orthosis in the last month
* Disorder of cognition or cooperation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Mouth Handicap in Systemic Sclerosis Questionnaire (MHISS) | at first day and second week change
  Mouth Handicap in Systemic Sclerosis Questionnaire (MHISS): This is a self-reported scale specific to the disease that questions oral involvement in systemic sclerosis. It consists of 12 items that evaluate features such as mouth opening, chewing, tooth structure, lip structure, dry mouth, fluent speech, and facial appearance. It is answered according to the five-point Likert system: 0: Never, 1: Rarely, 2: Sometimes, 3: Frequently, 4: Always. The higher the total score, the higher the severity of the problem.

SECONDARY OUTCOMES:
Scleroderma Health Assessment Questionnaire (SHAQ) | at first day
  Scleroderma Health Assessment Questionnaire (SHAQ): The SHAQ includes 5 visual analog scale questions that question Raynaud's phenomenon, digital ulcer, gastrointestinal and pulmonary respiratory symptoms, as well as the patient's overall disease severity. In addition, there are 20 questions (HAQ) evaluating the functional competence level of the patient. Each question is between 0-3 points (0: no difficulty and 3: can not). In the scoring of the sections, the highest score among the items constituting that section is accepted as the section score. The score of each category is summed and divided by the total number of categories, 8 to obtain the SHAQ disability score.
Oral Health Impact Profile (OHIP-14) | at first day
  It is a self-report scale that questions the proportion of individuals experiencing oral health problems. Likert response system; 0: None, 1: Rarely, 2: Sometimes, 3: Often, 4: Very often. The evaluation shows the total score of the participants' responses to each item, while OHIP-14 A (additive) shows the number of responses that a participant gave as 2 (sometimes) and 3 (often) in 14 items. The increase in the total score indicates that the severity of the problem increases and quality of life decreases.
Eating Assessment Tool (EAT-10) | at first day
  It is a single factor scale used to evaluate the severity and change of dysphagia symptoms. It consists of ten items. Each item is scored from 0 to 4. The total score ranges from 0 to 40. The scale is considered to be abnormal 3 points or more.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA CIVI KARAASLAN, MSc, Principal Investigator — Research Assistant
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mouthon L, Rannou F, Berezne A, Pagnoux C, Arene JP, Fois E, Cabane J, Guillevin L, Revel M, Fermanian J, Poiraudeau S. Development and validation of a scale for mouth handicap in systemic sclerosis: the Mouth Handicap in Systemic Sclerosis scale. Ann Rheum Dis. 2007 Dec;66(12):1651-5. doi: 10.1136/ard.2007.070532. Epub 2007 May 14. PMID 17502364
- [Background] Maddali Bongi S, Del Rosso A, Miniati I, Galluccio F, Landi G, Tai G, Matucci-Cerinic M. The Italian version of the Mouth Handicap in Systemic Sclerosis scale (MHISS) is valid, reliable and useful in assessing oral health-related quality of life (OHRQoL) in systemic sclerosis (SSc) patients. Rheumatol Int. 2012 Sep;32(9):2785-90. doi: 10.1007/s00296-011-2049-x. Epub 2011 Aug 17. PMID 21847653
- [Background] Schouffoer AA, Strijbos E, Schuerwegh AJ, Mouthon L, Vliet Vlieland TP. Translation, cross-cultural adaptation, and validation of the Mouth Handicap in Systemic Sclerosis questionnaire (MHISS) into the Dutch language. Clin Rheumatol. 2013 Nov;32(11):1649-55. doi: 10.1007/s10067-013-2321-4. Epub 2013 Jul 24. PMID 23881437
- [Background] Scardina GA, Messina P. Systemic sclerosis: description and diagnostic role of the oral phenomena. Gen Dent. 2004 Jan-Feb;52(1):42-7. PMID 15055670
- [Background] Naylor WP, Douglass CW, Mix E. The nonsurgical treatment of microstomia in scleroderma: a pilot study. Oral Surg Oral Med Oral Pathol. 1984 May;57(5):508-11. doi: 10.1016/0030-4220(84)90309-8. PMID 6587299